CLINICAL TRIAL: NCT05904691
Title: Safety and Tolerability of Single Ascending Doses and Multiple Repeat Doses of OCU-10-C-110 for Injection in Study Participants With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: Safety and Tolerability of OCU-10-C-110 for Injection in Subjects With Neovascular Age-related Macular Degeneration
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ocugenix Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCU-10-C-110-CS101
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD)
Keywords: neovascular age-related macular degeneration; intravitreal
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label, two-part safety assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A - Dose 1 (Experimental)
  Interventions: Drug: OCU-10-C-110 for Injection
- Cohort A - Dose 2 (Experimental)
  Interventions: Drug: OCU-10-C-110 for Injection
- Cohort A - Dose 3 (Experimental)
  Interventions: Drug: OCU-10-C-110 for Injection
- Cohort B - Dose TBD (Experimental)
  Interventions: Drug: OCU-10-C-110 for Injection

INTERVENTIONS:
Drug: OCU-10-C-110 for Injection — OCU-10-C-110 for Injection in one of 3 doses

SUMMARY:
Multi-center, open-label, two-part safety assessment following administration of single ascending doses and repeat administration of the HTD of OCU-10-C-110 for Injection in the study eye of participants with nAMD

DETAILED DESCRIPTION:
In Part A, subjects will receive a single intravitreal dose in a single eye of the drug product. Dose will be escalated in 3 successive cohorts, pending safety. In Part B, subjects will receive 3 treatments in a single eye of drug product at 4 week intervals of the maximally tolerated dose, with an additional 4 weeks of observation for safety. .

ELIGIBILITY:
Inclusion Criteria:

1. Angiographically documented active choroidal neovascular (CNV) lesion (i.e., leakage on fluorescein angiography or subretinal, intraretinal, or sub-retinal pigment epithelium [sub-RPE] fluid on spectral domain optical coherence tomography [SD-OCT]) secondary to age-related macular degeneration (AMD), within the previous 10 weeks
2. Subjects must have received, 7 to 14 days prior to the Baseline Visit, an intravitreal injection in the study eye of an anti-vascular endothelial growth factor (VEGF) ocular therapeutic approved for use in the United States

Exclusion Criteria:

1. History or current evidence of a medical condition (systemic or ophthalmic disease, metabolic dysfunction, physical examination finding or clinical laboratory finding) that may, in the opinion of the investigator, preclude the safe administration of the study medication, adherence to the scheduled study visits, or safe participation in the study or affect the results of the study (e.g., unstable or progressive cardiovascular, cerebral vascular, pulmonary, Parkinson's, liver or renal disease, depression, cancer, or dementia)
2. History or evidence of the following surgeries/procedures in the study eye:

   1. Submacular surgery
   2. Vitrectomy
   3. Retinal detachment or retinal tear
   4. Incisional glaucoma surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Ocular safety - AE | Cohort A - 8 weeks; Cohort B - 12 weeks
  Number of Adverse events

SECONDARY OUTCOMES:
Systemic safety - AE | Cohort A - 8 weeks; Cohort B - 12 weeks
  Number of Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldberg, MD, Study Director — Lexitas Pharma
Locations (3):
- United States (3):
  - Raj K. Maturi, M.D., P.C., Carmel, Indiana
  - Retina Research Institute of Texas, Abilene, Texas
  - Strategic Clinical Research Group LLC, Willow Park, Texas

IPD SHARING:
Plan to Share IPD: No
No sharing plans for this Phase 1 study at this time.